CLINICAL TRIAL: NCT02018588
Title: Tryptophan Requirement of Healthy School Age Children Determined by the Indicator Amino Acid Oxidation Method
Brief Title: Tryptophan Requirement of Healthy School Age Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Dr. Paul Pencharz, Professor of Paediatrics and Nutritional Sciences (Emeritus) University of Toronto, Senior Scientist Research Institute, The Hospital for Sick Children, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0019850580T
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: requirements; amino acid; tryptophan
MeSH Terms: interventions — Tryptophan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tryptophan intake (Experimental): Graded levels of tryptophan will be given to each subject on different study days around the anticipated breakpoint.
  Interventions: Dietary Supplement: tryptophan

INTERVENTIONS:
Dietary Supplement: tryptophan — graded levels of tryptophan will be given to each subject

SUMMARY:
Our objective is to determine the requirement for the amino acid tryptophan in school age children using the indicator amino acid technique.

DETAILED DESCRIPTION:
Seven healthy children will participate in the study. The children will participate as an outpatient basis with study days carried out in the Physiological Research Unit at the Hospital of Sick Children, Toronto, Canada. Inclusion criteria include: being healthy, not taking any medications, no recent weight changes, no history of significant illness, willing to participate in the study. Exclusion criteria were the presence of illness, significant weight change, not acceptance of the diet. Prior to enrolment, each subject will have to fill 3 days food record form to ensure his or her normal dietary behavior. The study will be explained to subjects and their parents/guardians, benefits and potential risks will be explained as well and written assent, from the children, and consent from parents will be obtained. Subjects will receive financial compensations. Each subject will receive compensation for participation. Each parent/guardian will be reimbursed for the transpiration/parking expenses and a meal each study day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children age 6-10 inclusive

Exclusion Criteria:

* significant recent illness

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2013-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Requirement of tryptophan in school age children | 4 hours
  By collection of stable isotope labeled CO2 from the indicator amino acid phenylalanine in response to different intake levels of tryptophan we will be able to determine tryptophan requirements.

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Pencharz, MD, PhD, Principal Investigator — The Hospital for Sick Children, Toronto, Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Mokbel A, Courtney-Martin G, Elango R, Ball RO, Pencharz PB, Tomlinson C. Tryptophan Requirement in School-Age Children Determined by the Indicator Amino Acid Oxidation Method is Similar to Current Recommendations. J Nutr. 2019 Feb 1;149(2):280-285. doi: 10.1093/jn/nxy250. PMID 30753549